CLINICAL TRIAL: NCT04038021
Title: Phosphatidylethanol-Based Contingency Management to Reduce Alcohol Use and Improve Housing Outcomes
Brief Title: Phosphatidylethanol-Based Contingency Management for Housing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington State University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Michael McDonell, Associate Professor, Washington State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17752; R21AA027045-01A1 (NIH)
Record Dates: First submitted 2019-07-24; First posted 2019-07-30 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2023-04

CONDITIONS: Alcohol Use Disorder
Keywords: Unstably Housed; Homeless
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PEth-based CM (Experimental): PEth-based CM participants will receive gift cards (starting at $30) each time they submit a blood spot sample (via finger prick ) with a negative alcohol result. They will receive an additional $5 (building on the previous amount) for each additional negative alcohol result in a row. There is a cap at $100 for each negative result.
  Interventions: Behavioral: Phosphatidylethanol-based Contingency Management
- Non-contingent Control (Active Comparator): Non-contingent control participants will receive gift cards each visit if they provide a pinprick blood sample regardless of whether the results are positive or negative for alcohol. Their level of reinforcement (amount in gift cards) will be equal to the average weekly CM earnings from the previous month.
  Interventions: Behavioral: Non-Contingent Control

INTERVENTIONS:
Behavioral: Phosphatidylethanol-based Contingency Management — In CM, tangible reinforcers are provided after individuals demonstrate biochemically verified abstinence of various substances. CM is associated with increased abstinence from illicit drugs, nicotine, and alcohol and is the most powerful psychosocial treatment for initiating abstinence of these substances. When participants submit a negative result for alcohol (via blood phosphatidylethanol biomarkers), the subject will receive rewards (gift cards). In contrast, they will not receive rewards when their samples test positive for alcohol.
  Other Names: Contingency Management (CM)
  Arms: PEth-based CM
Behavioral: Non-Contingent Control — In the non-contingent control intervention, participants will receive rewards (gift cards) regardless of the alcohol biomarker results in their samples. Once the samples have been received, the subjects will receive reinforcers that is consistent with the average from the CM group's earnings.
  Arms: Non-contingent Control

SUMMARY:
The investigators will evaluate the efficacy of contingency management (CM) in reducing alcohol use in individuals experiencing unstable housing but who are currently housed in shelters. Participants will be 20-30 adults diagnosed with alcohol use disorder (AUD) and has a history or unstable housing or literal homelessness in the last year but is currently receiving housing through Catholic Charities Spokane or other locations. Individuals who demonstrate AUD and have measurable PEth >ng/mL at the baseline visit will be randomized to receive Phosphatidylethanol-based CM treatment or non-contigent treatment.

DETAILED DESCRIPTION:
The objective of this study is to determine whether CM intervention improves outcomes in the unstably housed population using alcohol biomarker phosphatidylethanol (PEth) and ethyl glucuronide (EtG) to test alcohol abstinence. In CM, participants receive tangible rewards for demonstrating drug abstinence while non-contingent intervention receive the rewards regardless of PEth and EtG results for alcohol.

The investigators propose to examine whether CM intervention, to reduce alcohol use to abstinence, is a feasible and acceptable treatment in supported housing. Additionally, this study will assess group differences (between PEth-based CM and non-contingent control) in alcohol abstinence, as assessed by PEth, EtG, and self-report. Characterization of group differences in housing status and other alcohol associated harms (e.g., physical and mental health, medical care, and incarceration) will also be analyzed.

A total of 20-30 participants receiving treatment as usual through Catholic Charities Spokane or other locations in the Pacific and Mountain Time Zones will take part. Participants with AUD and have PEth biomarker results above >20 ng/mL, which indicates regular alcohol usage will be randomized to

1. 6 months of PEth-based CM for submitting alcohol-abstinent PEth results of 16:0/18:1 which is associated with abstinence in the past week, which is <20 ng/ml PEth biomarker in the blood when abstinent for 14-28 days. Urine EtG results will be analyzed to verify PEth result findings,
2. 6 months of non-contingent control for submitting samples each week for the first 4 weeks then every 2 weeks for 4 weeks and then every 4 weeks until week 26. Control participants receive reinforcers regardless of the results of their PEth results. The primary outcomes will assess acceptability measured by attrition, Client Satisfaction Questionnaire-8 and qualitative interviews at weeks 4, 12, and 26. Other primary outcomes include assessment of the effectiveness of PEth-based CM on reducing alcohol use to abstinence and housing status.

The investigators will also be examining group differences in secondary outcomes including self-reported abstinence and heavy drinking assessed by the alcohol timeline follow back and urine EtG analyses. Other secondary outcomes include a) Addiction Severity Index Lite which assesses impact of alcohol us on psychiatric, legal, medical and family functioning, b) self-reported drug use and its severity.

ELIGIBILITY:
Inclusion Criteria:

1. Two heavy drinking episodes (Assigned Male at Birth > 4 standard drinks (SDs), Assigned Female at Birth > 3 SDs) in the prior 14 days OR >14 drinks in the past 2 weeks, confirmed by a PEth level >=20 ng/ml
2. DSM-5 diagnosis of a current Alcohol Use Disorder (AUD) as assessed by the Structured Clinical Interview for Diagnostic and Statistical Manual 5 (DSM-5);
3. Age >=18 years;
4. Currently housed at Catholic Charities Spokane or other locations in the Pacific and Mountain time zones; and
5. Previously, literally homeless or unstably housed (e.g., couch surfing) for > 1 month

Exclusion Criteria:

1. Current diagnosis of substance use disorder (other than AUD and tobacco), severe;
2. Inability to provide informed consent based on the MacArthur Competence Assessment Tool for Clinical Research (MacCAT-CR) and/or age over 65 and Inability to provide informed consent based on the mini-Montreal Cognitive Assessment (mini-MoCA);
3. Alcohol withdrawal-related seizure or hospitalization in prior 12 months; and
4. Psychiatrically or medically unsafe to participate, as assessed by the PI.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2020-01-13 (Actual); Primary Completion 2022-08-23 (Actual); Study Completion 2022-10-27 (Actual)

PRIMARY OUTCOMES:
Rate of Attrition to measure acceptability of PEth-based CM Intervention | 26 weeks of treatment (repeated measure) through study completion
  Tolerability of PEth-based CM procedures (pinprick blood sample) measured by attendance, or attrition, with CM noted as acceptable if attrition is less than or equal to 30%. Attrition will be defined as 1 month of no contact with study team.
Acceptability of PEth-based CM: Client Satisfaction Questionnaire-8 | Weeks 4, 8, 12, 16, 20, and 26; repeated measure to assess change in satisfaction through study completion
  Administration of Client Satisfaction Questionnaire-8, a brief measure of client satisfaction that has been validated in addiction treatment. The scale ranges from 1 to 4 with 4 indicating higher satisfaction. Total scores therefore range from 8 (least satisfaction) to 32 (highest satisfaction).
Qualitative interviews to assess satisfaction, feasibility and acceptability of PEth-based CM Intervention using Theory Domains Framework (TDF) | Weeks 4, 12, and 26; repeated measure to assess change in satisfaction, feasibility, and tolerability through study completion
  Assessed by TDF to encode interviews to provide comprehensive, theory-informed data to identify determinants of satisfaction, feasibility and acceptability of intervention
Incidence of alcohol abstinence assessed by PEth biomarker | Weeks 1, 2, 3, 4, 6, 8, 10, 12, 16, 20, 24, and 26; repeated measure to assess change through study completion
  Efficacy of PEth-based CM in reduction of alcohol consumption to abstinence assessed by measurement of PEth in blood samples. PEth biomarker assessed at 16:0/18:1 for 7 days or < 20 ng/ml which is consistent with 14-28 days of abstinence
Efficacy of PEth-based CM in Stabilization of Housing Status | Weeks 1, 4, 8, 12, 16, 20, and 26; repeated measure to assess change of housing through study completion
  Measured by self-report of housing status using the Residential Timeline Follow Back; includes number of days stably housed, temporarily housed, institutionally housed or literally homeless. Residential Timeline Follow Back classifies location description of housing into literal homelessness, institutional housing, temporary housing, or stable housing.

SECONDARY OUTCOMES:
Self-Reported Alcohol Usage | 26 weeks of treatment (repeated measure) through study completion
  Days self-reported abstinence, drinking or heavy drinking measured by the Alcohol Timeline Follow Back
Alcohol Usage as measured by Urine Ethyl Glucuronide (uEtG) | 26 weeks of treatment (repeated measure) through study completion
  uEtG collected and measured to determine alcohol usage in last 1-4 days; uEtG greater or equal to 300 ng/ml is identified as recent drinking occurrence
The Addiction Severity Index Lite | Weeks 1, 4, 8, 12, 16, 20, and 26 (repeated measure) through study completion
  Assesses alcohol use on psychiatry, legal, medical, and family functioning, as well as self-reported drug use and its severity. Scale ranges from 0 (no craving at all) to 4 (extreme cravings)

OTHER OUTCOMES:
Short-Form Health Survey-12 | Weeks 4, 8, 12, 16, 20, and 26 (repeated measure) through study completion
  Measures mental and physical functioning and overall health-related quality of life. The scale for health includes: poor, fair, good, very good, and excellent. The pain interference scale includes: not at all, a little bit, moderately, quite a bit, and extremely.
Non-Study Resource Form for Medical and Criminal Justice Utilization | Weeks 4, 8, 12, 16, 20, and 26 through study completion
  Measures outpatient addiction, mental health, primary care, and vocational services, as well as the emergency department, inpatient psychiatric, and medical hospitalizations, detox admissions, residential addiction treatment, arrests and incarcerations.
Substance Use Test | 26 weeks of treatment (repeated measure) through study completion
  Urine samples will be tested for opioids, amphetamine, methamphetamine, cocaine, and cannabis with E-Z split (type of urine analysis cup) point-of-care immunoassays
Cigarette Consumption | 26 weeks of treatment (repeated measure) through study completion
  Assessed with the Cigarette Timeline Follow Back to measure smoking and other nicotine use
Cognitive Functioning | Week 1 and 26 (repeated measure) through study completion
  Using a battery of cognitive tests from Test My Brain
Fagerstrom Test for Nicotine Dependence | 26 weeks of treatment (repeated measure) through study completion
  Assesses an individual's dependence on nicotine; score total range from 0 to 10 with 0 being no dependence and 10 being most intense physical dependence on nicotine
Alcohol-Related Incentive Salience | Weeks 1, 4, 8, 12, 16, 20, and 26 (repeated measure) through study completion
  Self-rating instrument that provides a total and two subscale scores that measure some cognitive aspects of alcohol cravings
Stages of Change Readiness and Treatment Eagerness Scale (SOCRATES) | Weeks 1, 4, 8, 12, 16, 20, and 26 (repeated measure) through study completion
  19-item scale measuring an individual's eagerness to change drinking habits; each item has a score of 1 (strongly disagree) , 2 (disagree), 3 (not sure/undecided), 4 (agree), and 5 (strongly agree). There are three sub-scales for recognition, ambivalence, and taking steps in relation to drinking. The higher the score for each sub-scale indicate acknowledgement of drinking problem, uncertainty of control over drinking, and changing habits around drinking, respectively. Lower scores indicate denial of alcohol being a problem, not wondering about control of drinking, and not taking steps to change drinking, respectively.
Rate of Adverse Events | 26 weeks of treatment (repeated measure) through study completion
  Risks related to suicidality, dangerous alcohol use and withdrawal symptoms will be assessed
Emotional Functioning - Depression | Weeks 1, 4, 8, 12, 16, 20, and 26 (repeated measure) through study completion
  A questionnaire measuring the severity of depression (PHQ-9). PQQ-9 is scored on a 4 point scale: 1 (not at all), 2 (several days), 3 (more than half the days), and 4 (nearly every day).
Emotional Functioning - Anxiety | Weeks 1, 4, 8, 12, 16, 20, and 26 (repeated measure) through study completion
  A questionnaire measuring the severity of anxiety (GAD-7). GAD-7 is scored on a 4 point scale: 1 (not at all), 2 (several days), 3 (more than half the days), and 4 (nearly every day).
Emotional Functioning - Stress | Weeks 1, 4, 8, 12, 16, 20, and 26 (repeated measure) through study completion
  A questionnaire measuring the severity of stress (PSS). The PSS is scored on a 5 point scale: 0 (Never), 1 (Almost Never), 2 (Sometimes), 3 (Fairly Often), 4 (Very Often)

CONTACTS AND LOCATIONS:
Overall Officials: Michael G McDonell, PhD, Principal Investigator — Washington State University
Locations (1):
- Catholic Charities of Eastern Washington, Spokane, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jett JD, Beck R, Tyutyunnyk D, Sanchez J, Weeks DL, Javors MA, Hill-Kapturczak N, Lopez-Cruzan M, Kriegel L, Ginsburg BC, Cabassa L, McDonell MG. Feasibility of a telehealth-based contingency management intervention for alcohol use disorders using the phosphatidylethanol (PEth) 16:0/18:1 alcohol biomarker: a pilot randomized trial. Am J Drug Alcohol Abuse. 2024 Mar 3;50(2):162-172. doi: 10.1080/00952990.2023.2283691. Epub 2024 Jan 29. PMID 38284925